CLINICAL TRIAL: NCT06615180
Title: Evaluating the Effectiveness of a New Curriculum for Transcultural Nursing Education: a Mixed-method Study
Brief Title: Evaluating the Effectiveness of a New Curriculum for Transcultural Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Hasan Kalyoncu University (Other); Giresun University (Other)
Responsible Party: Principal Investigator, BETÜL TOSUN, PhD, Aassoc. Prof, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/07
Record Dates: First submitted 2024-09-18; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2022-02

CONDITIONS: Nursing Education; Cultural Competence; Cultural Sensitivity
Keywords: Nursing students; transcultural nursing; nursing education; cultural competence; cultural sensitivity; metaphor analysis

STUDY DESIGN:
Intervention Model Description: This international curriculum was developed with researchers from seven institutions and five countries (Turkey, Spain, Czech Republic, Belgium, Slovenia, and Hungary). The transcultural nursing course, which implemented 25 hours in a one-semester elective course, had 8 hours of theoretical training and 17 hours of practical training in two nursing departments in Turkiye . The course has 3 ETCSs (a 75 h workload for the students). This elective, the Transcultural Nursing Course was chosen by 5th-semester BSc nursing students.
  The aim of the course was To develop/promote awareness of culture-based care; it is aimed that at the end of this course, students would be capable of evaluating individuals, families, and communities in a proper and evidence-based manner, and they would be competent to plan, implement and evaluate culture-based nursing care. Learning outputs were prepared based on culture care theory by Madeleine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcultural Nursing Course (new curriculum) (Other): The Transcultural Nursing Course is a 25-hour elective designed to promote cultural competence in nursing students. It consists of 8 hours of theoretical instruction and 17 hours of practical training. The course is based on Madeleine Leininger's Culture Care Theory and incorporates models such as the Purnell, Campinha-Bacote, and Papadopoulos Models of Cultural Competence. It is aimed at enabling students to provide culturally appropriate nursing care for individuals, families, and communities.
  Interventions: Behavioral: Transcultural Nursing Course (new curriculum)

INTERVENTIONS:
Behavioral: Transcultural Nursing Course (new curriculum) — Multinational Collaboration: Developed with input from institutions across five countries, ensuring a broad, international perspective on transcultural nursing.
  Comprehensive Theoretical Framework: Integrates multiple cultural competence models (Purnell, Campinha-Bacote, Papadopoulos) with Leininger's Culture Care Theory, offering a thorough approach.
  Extensive Practical Training: Includes 17 hours of hands-on experience, featuring hospital visits and interactions with healthcare professionals.
  Interactive Learning Methods: Combines role-playing, reflective essays, and cultural activities (e.g., traditional clothing, dances) for dynamic, multimodal education.
  Peer Education: Incorporates peer education and evaluation, enhancing collaborative learning and critical thinking.
  Standardized Materials: Educational materials and teaching methods are standardized across institutions to ensure consistency and quality in instruction.
  Other Names: Culture-Based Nursing Care Education

SUMMARY:
In recent years, limited studies have evaluated the development of cultural awareness, sensitivity, skills, communication, and competence among nursing students using different models and curricula. This study aims to evaluate the effectiveness of a new internationally developed curriculum for transcultural nursing education. This mixed methods study was conducted on nursing students (n=83) who attended a transcultural nursing course from 2021-2022 during the fall semester.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Volunteering to participate in the research
* Being enrolled in the Transcultural Nursing Course in the fall semester 2021-2022

Exclusion Criteria:

* Not meeting the criteria for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Better and Effective Nursing Education for Improving Transcultural Nursing Skills Cultural Competence and Cultural Sensitivity (BENEFITS-CCCS) Scale | At baseline, 15 minutes before the first class, students were informed about the BENEFITS-CCC Scale, and the survey was administered. The scale was re-applied 15 minutes before the final class ended, following the completion of the 14-week curriculum
  This scale was developed by researchers from Belgium, the Czech Republic, Hungary, Slovenia, Spain, and Türkiye in the project Better and Effective Nursing Education for Improving Transcultural Nursing Skills (BENEFITS) to evaluate the effectiveness of cultural competence training in nursing students. The scale has 26 items across five subdimensions: Respect for Cultural Diversity (6 items), Culturally Sensitive Communication (4 items), Achieving Cultural Competence (3 items), Challenges and Barriers in Providing Culturally Competent Care (5 items), and Perceived Meaning of Cultural Care (8 items). Items are scored on a 7-point Likert scale (1 for Definitely Disagree to 7 for Definitely Agree). The possible total score ranges from 26 to 182. The scale Cronbachs alpha is 0.82.

OTHER OUTCOMES:
Metaphor Analysis Tool for Assessing Transcultural Nursing Experiences | Post-course assessment at the end of the semester (14 week). Students submitted their answers to the questions in essay form in the 15th week.
  Unit of Measure:
  Qualitative themes derived from metaphorical expressions related to experiences with patients and teammates from diverse backgrounds.
  Measurement Tool:
  A qualitative questionnaire prompting nursing students to complete the following statements:
  1. Caring for patients with different religions, languages, cultures, or lifestyles is like … because …
  2. Working with teammates having different religions, languages, cultures, or lifestyles is like … because …
  3. A culturally sufficient care environment is like … because …
  4. This transcultural nursing course is like … because …
  Data Analysis Process:
  Data were analyzed thematically, which involved coding the content into categories, defining themes, and interpreting results. Feedback was solicited from participants to ensure data validity, with three researchers reviewing the data and an expert opinion sought for reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Tosun, RN, PhD, Assoc. Prof., Study Director — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Giresun Üniversity, Giresun, Merkez
  - Hasan Kalyoncu University, Gaziantep, şehitkamil

IPD SHARING:
Plan to Share IPD: No
Individual data will be protected and presented in an anonymized form. The data will be used solely for scientific purposes, and informed consent from participants has been obtained under these conditions. Participant privacy and data security are prioritized. IPD sharing will be conducted in compliance with ethical and legal requirements. Measures will be taken to ensure data security and to grant access only to authorized researchers.